CLINICAL TRIAL: NCT00232492
Title: Effect of Racemic Ketamine on Pain in Females and Males After Surgical Removal of Third Molars
Brief Title: Ketamine on Acute Pain in Females and Males
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ullevaal University Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Professor Lasse A. Skoglund, Section of Dental Pharmacology and Pharmacotherapy, University of Oslo, Norway
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DOK-015
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2008-04

CONDITIONS: Mouth and Tooth Diseases; Tooth, Impacted
Keywords: Wisdom; Tooth; Teeth; Third; Molar
MeSH Terms: conditions — Stomatognathic Diseases; Tooth, Impacted

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- Placebo males (Placebo Comparator): Saline physiological placebo males
  Interventions: Drug: Placebo males
- Ketamine 0,1 mg/kg males (Active Comparator): 0,1 mg/kg ketamine males
  Interventions: Drug: Ketamine 0,1 mg/kg males
- Ketamine 0,3 mg/kg males (Active Comparator): 0,3 mg/kg ketamine males
  Interventions: Drug: Ketamine 0,3 mg/kg males
- Ketamine 0,5 mg/kg males (Active Comparator): 0,5 mg/kg ketamine males
  Interventions: Drug: Ketamine 0,5 mg/kg males
- Placebo females (Placebo Comparator): Saline physiological as placebo females
  Interventions: Drug: Placebo females
- Ketamine 0.1 mg/kg females (Active Comparator): 0,1 mg/kg ketamine females
  Interventions: Drug: Ketamine 0,1 mg/kg females
- Ketamine 0,3 mg/kg females (Active Comparator): 0,3 mg/kg ketamine females
  Interventions: Drug: Ketamine 0,3 mg/kg females
- Ketamine 0,5 mg/kg females (Active Comparator): 0,5 mg/kg ketamine females
  Interventions: Drug: Ketamine 0,5 mg/kg females

INTERVENTIONS:
Drug: Placebo males — Intravenous saline bolus (Placebo-control) males
  Other Names: saline physiological 5 ml
  Arms: Placebo males
Drug: Ketamine 0,1 mg/kg males — 0,1 mg/kg ketamine iv bolus males
  Other Names: Ketalar ATC-nr.: N01A X03
  Arms: Ketamine 0,1 mg/kg males
Drug: Ketamine 0,3 mg/kg males — 0,3 mg/kg ketamine iv bolus males
  Other Names: Ketalar ATC-nr.: N01A X03
  Arms: Ketamine 0,3 mg/kg males
Drug: Ketamine 0,5 mg/kg males — 0,5 mg/kg ketamine iv bolus males
  Other Names: Ketalar ATC-nr.: N01A X03
  Arms: Ketamine 0,5 mg/kg males
Drug: Placebo females — Intravenous saline bolus (Placebo-control) females
  Other Names: Saline physiological 5 ml
  Arms: Placebo females
Drug: Ketamine 0,1 mg/kg females — 0,1 mg/kg iv bolus ketamine females
  Other Names: Ketalar ATC-nr.: N01A X03
  Arms: Ketamine 0.1 mg/kg females
Drug: Ketamine 0,3 mg/kg females — 0,3 mg/kg iv bolus ketamine females
  Other Names: Ketalar ATC-nr.: N01A X03
  Arms: Ketamine 0,3 mg/kg females
Drug: Ketamine 0,5 mg/kg females — 0,5 mg/kg iv bolus ketamine females
  Other Names: Ketalar ATC-nr.: N01A X03
  Arms: Ketamine 0,5 mg/kg females

SUMMARY:
The purpose of the study is to determine whether equal subanesthetic doses of racemic ketamine is equally effective on females and males after surgical removal of third molars

DETAILED DESCRIPTION:
Ketamine is assumed to be a NMDA receptor antagonist which provides analgesia from acute postoperative pain(and other types of pain) subanesthetic doses. Gender differences in ketamine analgesia are not known. This placebo-controlled,randomised, parallel group study investigates the analgesic dose-response effect of ketamine in subanesthetic doses in female and male patients following surgical removal of third molars.

Comparisons: Placebo and ketamine in females and males.

ELIGIBILITY:
Inclusion Criteria:

* Indication for removal of third molar
* Between 20 and 30 years of age
* ASA Class 1

Exclusion Criteria:

* Psychiatric family (father/mother) or own anamnestic history
* Hypersensitivity towards NSAIDS or other rescue analgesics
* Verified or suspected pregnancy
* Lactating females
* Surgery lasting over 60 min

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2005-01; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Sum pain NRS | 60 min

SECONDARY OUTCOMES:
Several subjective variables assessing psychotomimetic effects | 0, 15, 60

CONTACTS AND LOCATIONS:
Overall Officials: Lasse A Skoglund, DDS, PhD, Study Chair — Section of Dental Pharmacology and Pharmacotherapy, Faculty of Dentistry, POB 1119 Blindern, University of Oslo, N-0317 Oslo, Norway; Olav Hustveit, MD, Principal Investigator — Section of Dental Pharmacology and Pharmacotherapy, Faculty of Dentistry, POB 1119 Blindern, University of Oslo, N-0317 Oslo, Norway
Locations (1):
- Department of Oral and Maxillofacial Surgery, Ullevaal University Hospital, Oslo, Norway

REFERENCES:
- [Background] Oye I, Mathisen LC. The effect of CPP in neurogenic pain: inhibition of spinal or cortical NMDA receptors? Pain. 1993 Jun;53(3):358. doi: 10.1016/0304-3959(93)90234-G. No abstract available. PMID 8351166
- [Background] Øye I, Hustveit O, Maurset A, Ratti Moberg E, Paulsen O, Skoglund LA. The chiral forms of ketamine as probes for NMDA receptor functions in humans. In: NMDA receptor related agents: Biochemistry, pharmacology and behaviour. Kameyama T, Domino E (eds). NPP Books, Ann Arbor, 1991.